CLINICAL TRIAL: NCT05499338
Title: Motivation as a Strategy for Adherence to a Stretching Program for Basketball Players: a Pilot Study.
Brief Title: Motivation as a Strategy for Adherence to a Stretching Program for Basketball Players
Acronym: MOTBAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, CRISTINA ADILLÓN, Principal Investigator, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 123/2018_2
Record Dates: First submitted 2022-08-08; First posted 2022-08-12 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Motivation; Sports Physical Therapy; Muscle Tightness

STUDY DESIGN:
Intervention Model Description: Single-blind, randomized, controlled, experimental clinical trial.
Who Masked: Investigator
Masking Description: The investigators were blinded, so that the initial and final investigators did not know which group everyone belonged to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group received a lecture session explaining what stretching is, its advantages and the importance of stretching in injury prevention. The specific intervention programme was to be performed at least 3 days/week (after training) for 12 weeks. These were static, active stretches of the muscles of the lower back, psoas iliacus, quadriceps, adductors, gluteus, hamstrings, and sural triceps. For each muscle group, the stretch was held for 60 seconds, divided into 3 repetitions of 20 seconds. Between each repetition, we did not return to the initial position but sought a new barrier to the stretch which would provoke the sensations described above. The total time dedicated to stretching was approximately 15 minutes per session.
  Interventions: Procedure: Stretching program
- Control group (No Intervention): The control group performed the initial and final assessments and continued to perform their team's standard/habitual stretches. To record whether they performed the stretches prescribed by the club, the researchers went to the end of the training unknown sessions and recorded whether the players performed them or not.

INTERVENTIONS:
Procedure: Stretching program — The stretching programme was to be performed at least 3 days/week (after training) for 12 weeks. These were static, active stretches of the muscles of the lower back, psoas iliacus, quadriceps, adductors, gluteus, hamstrings, and sural triceps. The final stretching position was that which generated a sensation of moderate-intense tightness in the muscles, but without exceeding the pain threshold. For each muscle group, the stretch was held for 60 seconds, divided into 3 repetitions of 20 seconds. Between each repetition, we did not return to the initial position but sought a new barrier to the stretch which would provoke the sensations described above. The total time dedicated to stretching was approximately 15 minutes per session.
  Arms: Experimental group

SUMMARY:
Background: Basketball is considered a medium-high injury sport, because of the mechanisms of injury, which can be acute, by repetition mechanisms or by overload. An effective way to avoid muscle overload injuries is to perform an extensibility workout such as an analytical active stretching program. The objective of this study is to achieve adherence to a stretching program by motivating young basketball players.

Methods: Randomized experimental clinical trial controlled by a single blind person. 21 child players between 11 and 12 years, divided into intervention group (IG) and control group (CG). IG carries out a supervised static stretching program at the end of training 3 days/week for 12 weeks and CG has normally developed the standard stretches of their Basketball Club. The extensibility of various muscle groups was valued in both groups. In addition, motivation was valued by Sport Motivation Scale.

DETAILED DESCRIPTION:
The inclusion criteria were: to be between 12 and 13 years of age (both included), to be an active player at the time of selection, to sign the informed consent form and failure to meet the exclusion criteria. The exclusion criteria were: to have an injury at the time of selection and psychological and/or psychiatric illnesses. The main outcomes were: the adherence to a stretching program (monitoring calendars), the extensibility of the posterior musculature (fingertip-to-floor test), the adductor extensibility (sideways leg splits test), the gastrocnemius and soleus extensibility (weight-bearing lunge test through the Leg Motion system), the hamstring extensibility (goniometer with the passive straight leg raise and it was considerated shortening if it doesn't reach >80 degrees of elevation, the extensibility of the quadriceps (Ely test by a goniometer), the extensibility of the psoas (modified Thomas test using a goniometer).

ELIGIBILITY:
Inclusion Criteria:

* To be an active player at the time of selection, to sign the informed consent form, failure to meet the exclusion criteria.

Exclusion Criteria:

* To have an injury at the time of selection, psychological and/or psychiatric illnesses.

Ages: 12 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Extensibility of the posterior musculature (centimeters) | 1 year
  This was measured with the "Fingertip-to-Floor Test"
Adductor extensibility (centimeters) | 1 year
  It was measured with the Sideways Leg Splits test
Gastrocnemius and soleus extensibility (centimeters) | 1 year
  The Leg Motion System was used.
Hamstring extensibility (degrees) | 1 year
  The Passive Straight Leg Raise test was used, assessed qualitatively and quantitatively.
Extensibility of the quadriceps (degrees) | 1 year
  This was measured with the Ely Test
Extensibility of the psoas (degrees) | 1 year
  The Modified Thomas test was used, assessing the psoas qualitatively and quantitatively as well as indirectly the rectus femoris, the tensor fascia lata and the abductors.
Motivation | 1 year
  It was assessed using the Sport Motivation Scale, validated in Spanish. This scale allows an objective assessment of the intrinsic, extrinsic and non-motivational factors of why children participate in their sport. In addition, the researchers added two questions related to motivation and stretching, to check whether the participants had correctly understood the importance of stretching.
Adherence to the programme (percentage) | 1 year
  This was assessed by means of monitoring calendars. The purpose of these was for the athletes to place blue stickers on the days they did the stretches and red stickers on the days they did not do them, thus giving them visual biofeedback of their involvement with the stretches. Each calendar was valid for six weeks, so one was given out on the first week and the second one in the middle of the study, on the sixth week.

SECONDARY OUTCOMES:
Age | 1 year
  Years
Gender | 1 year
  Female or male
Height | 1 year
  Centimeters
Hypermobility | 1 year
  The Beighton Criteria were used.

CONTACTS AND LOCATIONS:
Locations (1):
- Federación Catalana de Baloncesto, Barcelona, Spain

REFERENCES:
- [Background] Cumps E, Verhagen E, Meeusen R. Prospective epidemiological study of basketball injuries during one competitive season: ankle sprains and overuse knee injuries. J Sports Sci Med. 2007 Jun 1;6(2):204-11. eCollection 2007. PMID 24149330
- [Background] Sainz de Baranda P, Ayala F. Chronic flexibility improvement after 12 week of stretching program utilizing the ACSM recommendations: hamstring flexibility. Int J Sports Med. 2010 Jun;31(6):389-96. doi: 10.1055/s-0030-1249082. Epub 2010 Mar 22. PMID 20309785
- [Background] Behm DG, Blazevich AJ, Kay AD, McHugh M. Acute effects of muscle stretching on physical performance, range of motion, and injury incidence in healthy active individuals: a systematic review. Appl Physiol Nutr Metab. 2016 Jan;41(1):1-11. doi: 10.1139/apnm-2015-0235. Epub 2015 Dec 8. PMID 26642915
- [Background] Bozic PR, Pazin NR, Berjan BB, Planic NM, Cuk ID. Evaluation of the field tests of flexibility of the lower extremity: reliability and the concurrent and factorial validity. J Strength Cond Res. 2010 Sep;24(9):2523-31. doi: 10.1519/JSC.0b013e3181def5e4. PMID 20802292
- [Background] Calatayud J, Martin F, Gargallo P, Garcia-Redondo J, Colado JC, Marin PJ. The validity and reliability of a new instrumented device for measuring ankle dorsiflexion range of motion. Int J Sports Phys Ther. 2015 Apr;10(2):197-202. PMID 25883868
- [Background] Ayala F, Sainz de Baranda P, De Ste Croix M, Santonja F. Comparison of active stretching technique in males with normal and limited hamstring flexibility. Phys Ther Sport. 2013 May;14(2):98-104. doi: 10.1016/j.ptsp.2012.03.013. Epub 2012 Sep 21. PMID 23007137